CLINICAL TRIAL: NCT05527418
Title: Safety, Tolerance and Antiretroviral Activity of Dasatinib: a Pilot Clinical Trial in Patients With Recent HIV-1 Infection
Acronym: DASAHIVCURE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eva Bonfill (Other)
Responsible Party: Sponsor-Investigator, Eva Bonfill, Clinical Research Manager, Institut d'Investigacions Biomèdiques August Pi i Sunyer
Organization: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-001288-26
Record Dates: First submitted 2022-08-03; First posted 2022-09-02 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Recent HIV-1 Infection
MeSH Terms: interventions — Dasatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dasatinib (Experimental): Dasatinib monotherapy (70 mg/day) will be given for 4 weeks. Antiretroviral therapy (ART) based on unboosted integrase inhibitors will be initiated at week 4 (S4) and dasatinib will be continued with ART until week 12.
  Interventions: Drug: Dasatinib
- Placebo (Placebo Comparator): Placebo monotherapy will be given for 4 weeks. Antiretroviral therapy (ART) based on unboosted integrase inhibitors will be initiated at week 4 (S4) and placebo will be continued with ART until week 12.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dasatinib — Dasatinib monotherapy 70 mg/day, during 16 weeks.
  Arms: Dasatinib
Drug: Placebo — Placebo during 16 weeks.
  Arms: Placebo

SUMMARY:
Study to evaluate the safety, tolerability and antiretroviral activity of a new therapeutic strategy, based on the administration of dasatinib, an ITK, in patients with recent (3-12 months) asymptomatic HIV-1 infection.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years.
* Documented asymptomatic HIV-1 infection of 3-12 months duration (all patients must have a positive Western blot, including the p31 band whose appearance indicates infection of more than 90 days duration).
* Not having received ART
* CD4 T-lymphocyte count> 350 / μl
* Patient giving written informed consent

Exclusion Criteria:

* Active HBV (HBsAg+ or DNA+) and/or HCV (RNA+) infection in screening.
* ALT> 2 UNL, glomerular filtration rate <70 mL / 1.73 m2, leukocytes <4000 / mm3, total lymphocyte count <1000 / mm3, platelets <100,000 / mm3 or Hg <12g / dL.
* Pregnancy or active breastfeeding
* Ongoing or previous pleural effusion
* Chronic obstructive pulmonary disease, bronchial asthma or recent chest trauma.
* History of gastrointestinal or other bleeding.
* Any concomitant treatment with potentially dangerous drug interaction with dasatinib.
* Any clinical condition, at the opinion of the investigator, contraindicating participation (for example,
* Active neoplastic disease, active concomitant infection, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerance of dasatinib with and without antiretroviral therapy, measured by number of AEs and SAEs | 52 weeks
  Measured by number of AEs and SAEs

SECONDARY OUTCOMES:
Antiretroviral capacity of dasatinib | at week 0 and 4
  Measured by quantification of plasma HIV-1 viral load during 4-week administration of dasatinib monotherapy.
Changes in the viral reservoirs of patients with recent HIV-1 infection induced by dasatinib administration. | at week 0, 4, 16 and 52
  Measured by changes in the viral reservoirs (integrated DNA, genetically intact virus, residual and induced viral replication and determination of integration sites)
Changes in markers of inflammation and immune activation induced by dasatinib administration. | at week 0, 4, 16 and 52
  Measured by changes in ultra-sensitive CRP, IL6, TNF alpha and CD4/CD8, CD25, CD69, CD38, HLA-DR+.
Changes in SAMHD1 phosphorylation levels and cytotoxic activity against HIV-1 induced by dasatinib. | at week 0, 4, 16 and 52
  Measured by NK phenotyping and in vitro replication inhibition tests.
Pharmacokinetic interactions of coadministration non-boosted integrase inhibitor-based antiretroviral therapy with dasatinib. | at week 1, 2, 3, 4, 8, 12, 16
  Measured by Cmax
Pharmacokinetic interactions of coadministration non-boosted integrase inhibitor-based antiretroviral therapy with dasatinib. | at week 1, 2, 3, 4, 8, 12, 16
  Measured by Cmin
Impact of dasatinib on markers of senescence | at week 0, 4, 16 and 52
  Measured by expression in PBLs of beta-galactosidase, Bcl-2, Histone H2A, p16 and CD87.

CONTACTS AND LOCATIONS:
Locations (1):
- Eva Bonfill, Barcelona, Spain